CLINICAL TRIAL: NCT06221904
Title: A The Effect of Simple Gymnastics Training for Parkinson's Patients in the Community: A Preliminary Study
Brief Title: The Effect of Simple Gymnastics Training for Parkinson's Patients in the Community
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-KY-0116
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The observation group (Experimental): The observation group is the only group.The elderly individuals will be arranged to undergo a continuous three-week (21 days) duration of Simple Gymnastics Training, with weekends off and training conducted only on weekdays, two sessions per day, each lasting 30 minutes. Each training session will be conducted approximately at 9.00 a.m. Apart from this,we require participants to only engage in daily activities and avoid strenuous and dangerous behaviors
  Interventions: Behavioral: Simple Gymnastics Training

INTERVENTIONS:
Behavioral: Simple Gymnastics Training — This is a simple gymnastics training that includes body swings and waist twists, as well as exercises targeting the joints in the arms and legs in various directions. It aims to help Parkinson's patients improve their physical mobility. Each training session lasts for 30 minutes, with low intensity and easy to stick to.

SUMMARY:
The goal of this clinical trial is to explore the impact of Simple Gymnastics Training on Limb motor function and mental health in Parkinson's Patients in the Community (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of Parkinson's Diseases among community-dwelling elderly individuals, and 2) the effects of Simple Gymnastics Training on Limb motor function and mental health in community-dwelling Parkinson's Patients. All patients are required to undergo a continuous three-week (21 days) Simple Gymnastics Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

DETAILED DESCRIPTION:
In the early stages of Parkinson's disease, many patients do not seek medical attention. The goal of this clinical trial is to explore the impact of Simple Gymnastics Training on Limb motor function and mental health in Parkinson's Patients in the Community (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of Parkinson's Diseases among community-dwelling elderly individuals, and 2) the effects of Simple Gymnastics Training on Limb motor function and mental health in community-dwelling Parkinson's Patients. All patients are required to undergo a continuous three-week (21 days) Simple Gymnastics Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years.
* Meeting the diagnostic criteria for Parkinson's disease developed by the Neurology Branch of the Chinese Medical Association in 2006.

Exclusion Criteria:

* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | day 1 and day 21
  The score of the Unified Parkinson's Disease Rating Scale ranges 0 to 199 points. This assessment tool includes items such as non-motor symptoms, motor function, activities of daily living, and complications, each with corresponding scoring criteria. Higher scores reflect more severe symptoms and functional impairments. The scale is a commonly used assessment tool that can be used to evaluate the severity and progression of Parkinson's disease, as well as the effectiveness of rehabilitation treatment.

SECONDARY OUTCOMES:
The Berg Balance Scale | day 1 and day 21
  The Berg Balance Scale is a scale used to assess balance ability. It is widely used in rehabilitation and research for patients with Parkinson's disease and other movement disorders.
  The scale consists of 14 items, each involving different balance tasks and actions such as standing, turning, walking, and more. Each item is scored based on the performance level, ranging from 0 to 4, with a maximum total score of 56. Higher scores indicate better balance ability.
Patient Health Questionnaire-9 | day 1 and day 21
  Patient Health Questionnaire-9 is a scale used to assess symptoms of depression, consisting of 9 items. Each item involves different aspects of depressive symptoms such as mood, sleep, appetite, etc. Each item is scored based on the frequency and severity of symptoms in the past two weeks, with a score range from 0 to 27. Higher scores indicate more severe symptoms. Patient Health Questionnaire-9 is widely used for screening and assessment of depression.
Generalized Anxiety Disorder-7 | day 1 and day 21
  Generalized Anxiety Disorder-7 is a scale used to assess symptoms of generalized anxiety disorder, consisting of 7 items. Each item involves different aspects of anxiety symptoms such as worry, tension, unease, etc. Each item is scored based on the frequency and severity of symptoms in the past two weeks, with a score range from 0 to 21. Higher scores indicate more severe symptoms. Generalized Anxiety Disorder-7 is widely used for screening and assessment of generalized anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Sumei Wang, Master, Study Director — Zhengzhou Tielu Hospital
Locations (1):
- Tielu Community, Kaifeng, Henan, China

IPD SHARING:
Plan to Share IPD: No